CLINICAL TRIAL: NCT05670626
Title: Correlation Between ICL Vault and Preoperative Refraction ( Spherical Equivalent) and Anterior Segment Parameters Measured by Optical Biometry and Scheimpflug Imaging
Brief Title: Correlation Between Preoperative Refraction and Anterior Segment Parameters With ICL Vault
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Nermine Said Aly Madkour, ophthalmology consultant, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MD-360-2021
Record Dates: First submitted 2022-12-11; First posted 2023-01-04 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Refractive Errors; Myopia; Myopic Astigmatism
Keywords: Refractive surgery; Phakic intraocular lens; ICL vault
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism | interventions — Refractive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- non comparative interventional study (Other): patients with high refractive error will do phakic ICL after preoperative assessment of anterior segments parameters and post-operative ICL vault will be measured using pentacam
  Interventions: Procedure: Refractive Surgery

INTERVENTIONS:
Procedure: Refractive Surgery — Phakic implantable contact lens ( ICL)

SUMMARY:
This prospective non-comparative interventional study aims to analyse the pre-operative factors affecting the range of optimal ICL vaulting. the main question is what is the correlation between age, gender, spherical equivalent, white to white, anterior chamber volume and depth and postoperative vault? participants will do preoperative investigations ( specular microscopy, pentacam and biometry ) then refractive surgery (ICL implantation) followed by follow-up visits to assess the post-operative ICL vault and visual outcome.

DETAILED DESCRIPTION:
Procedure: Refractive error correction by implantable contact lens ( ICL) will be preceded by a Preoperative assessment of the patient's anterior segment using specular Microscopy, pentacam and biometry and full ophthalmic examination.

Post-operatively, visual acuity evaluation, intraocular pressure, and anterior and posterior segments examination using a slit lamp will be done on days 1 and 3 and then repeated after 1 month and 6 months Assessment of ICL vault measurement using pentacam scheimpflug imaging after 1 and 6 months will be done then a correlation between the ICL vault and the patient's refractive error and preoperative anterior segments parameters will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Age:21 - 45 years old.
* High Myopia or Myopic astigmatism.
* Patients with stable preoperative refraction for the previous 12 months.
* Aqueous depth (ACD internal) = 2.8 mm or greater from the endothelial side using pentacam.
* Patients who are not fit for LASIK.
* No previous intraocular surgeries.

Exclusion Criteria:

* Patients with endothelial cell count < 2800 cells /mm2
* Patients with corneal opacities
* Patients with preoperative glaucoma, cataract, and retinal disease.
* Patients with any systemic diseases especially collagen diseases.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ICL vault size | 1 month
  assessment of ICL vault by scheimpflug image
ICL Vault size | 6 months
  assessment of ICL vault by scheimpflug image
Post Operative UCVA and BCVA | 1-3 days
  assessment of Post Operative visual acuity
Post Operative UCVA and BCVA | 1 month
  assessment of Post Operative visual acuity
Post Operative UCVA and BCVA | 6 months
  assessment of Post Operative visual acuity
Post Operative IOP | 1 - 3 days
  assessment of post operative intraocular pressure
Post Operative IOP | 1 month
  assessment of post operative intraocular pressure
Post Operative IOP | 6 month
  assessment of post operative intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Adel M Fathy, Prof. DR, Study Director — Faculty of medicine Kasr El Aini; Ramy R Fikry, Ass prof, Study Director — Faculty of medicine Kasr El Aini; Mohamed A Anis, Ass Prof, Study Director — Faculty of medicine Kasr El Aini
Locations (1):
- Alwatany Eye Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No